CLINICAL TRIAL: NCT03631121
Title: Effects of Replacing Lantus With Basalin on the Glycemic Variation in Patients
Brief Title: Effects of Replacing Lantus With Basalin on the Glycemic Variation in Patients With Type 2 Diabetes Mellitus
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KY20170904-01
Record Dates: First submitted 2018-08-12; First posted 2018-08-15 (Actual); Last update posted 2019-06-11 (Actual); Status verified 2018-08

CONDITIONS: Type2 Diabetes

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Basalin to Lantus (Experimental): the patients who are using Basalin treatment will use isodose of Lantus instead
  Interventions: Drug: Basalin to Lantus

INTERVENTIONS:
Drug: Basalin to Lantus — continuous glucose monitoring system will used twice when patients are using Basalin and Lantus respectively to assess glycemic variation.

SUMMARY:
The study will assess the glycemic variationusing continuous glucose monitoring system in type 2 diabetic patients with euglycemia control respectively when patients was treated with Basalin and one week after changing the insulin into Lantus.

DETAILED DESCRIPTION:
The participants will take continuous glucose monitoring system for 3 days when they change the insulin into Lantus after reach euglycemia control with Basalin treatment for one week.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with T2DM, which was defined bypublished Criteria of World Health Organization in 1999;
2. Patients were using Basalin with or without oral hypoglycemic drugs and having a stable dose of glargine for more than 3 month would be recruited into this study;
3. Patients had relatively constant diet and exercise in 2 month before the study.
4. Fasting blood glucose<6.1mmol/L, and postprandial (or random) blood glucose <14mmol/L

Exclusion Criteria:

1. Patients with severe cardiovascular diseases, such as stroke, transient ischemic attack, myocardial infarction, unstable angina, coronary artery bypass grafting, percutaneous coronary intervention, and heart failure;
2. Patients with severe infectious diseases;
3. Patients with acute complications of diabetes on admission, such as diabetic ketoacidosis, diabetic hyperosmolar nonketotic coma, and lactic acidosis;
4. Patients with history of psychiatric disorders and were unsuitable to use CGMS;
5. Any other situations that made patients unsuitable to participate in the study, such as alcoholism and drug abuse.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-08-15 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-07-30 (Estimated)

PRIMARY OUTCOMES:
Change of glycemic variation | Day 1-13
  The changes of glycemic variation before and after drug change

CONTACTS AND LOCATIONS:
Overall Officials: Ma Jianhua, Study Chair — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Nanjing First Hostital, Nanjing, Jiangsu, China